CLINICAL TRIAL: NCT01660087
Title: Diagnosis of Lung Cancer From Exhaled Breath With Silicon Biophotonic Device.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SERC/1121480001
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer
Keywords: Exhaled breath condensate (EBC) method; Volatile Organic Compounds (VOCs); Endobronchial Ultrasound (EBUS); Confocal Endoscopy; Exhaled alveolar gas
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Biophotonic platform for VOC detection — Multiplex detection of VOCs with high sensitivity and specificity using a novel biophotonic device.

SUMMARY:
The overall objective of this proposal is to develop a non-invasive, inexpensive and accurate device that detects VOCs in exhaled breath for lung cancer screening. Toward this goal, the team will design and fabricate a biophotonic platform consists of arrays of silicon micro-ring resonator sensors coated with polymers with different organic functionalities, in which each sensor is widely responsive to a variety of VOCs for the detection of lung cancer by means of breath testing. The team will identify signature VOCs as lung cancer biomarkers by comparison VOC contents between alveolar gas that directly sampled from the nodule or mass and exhaled breath using gas chromatography/ mass spectrometry.

The specific aims of this proposal are as followings:

Aim 1: To develop a biophotonic platform for the detection of VOCs

Aim 2: To achieve multiplex detection of VOCs with high sensitivity and specificity using a novel biophotonic device.

Aim 3: To evaluate the device as a lung cancer screening tool by testing both healthy and lung cancer breath samples

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths throughout the world and accounts for more than 1.2M new cases worldwide annually, making lung cancer one of the most serious public health problems in industrialized countries. Up to date there is no valid screening method for lung cancer. Thus it is often diagnosed at an advance stage when treatment is less effective, which consequantly leads to high mortality rate. However, with early diagnosis and treatment, the 5-year survival rate improves dramatically from 1% in stage 4, 20% in stage 3 to 70% in stage 1 disease. Therefore early diagnosis plays a pivotal role in improving survival for this otherwise uniformly fatal disease. In recently studies, it was found that some of the products of metabolism, called volatile organic comounds (VOCs), are carried in the breath and can serve as biomarkers. Cancer cells produce different types of VOCs than normal cells do. More importantly, these VOC markers can be found in exhaled breath for cancer stages 1 through 4.

Combining the strength of IME's in the biophotonics, the research groups at NUS in basic science and the NUH clinician's knowledge and expertise in lung cancer, this proposal is aiming to tackle the challenge of lung cancer screening by developing a non-invasive, inexpensive, and accurate sensor platform to detect VOCs in exhaled breath. The device will consists of arrays of silicon micro-ring resonator sensors coated with polymers with different organic functionalities, in which each sensor is widely responsive to a variety of VOCs. In this proposal, we plan to build a prototype device and test for the detection of VOCs in exhaled breath from healthy controls and lung cancer patients. The successful outcome of this proposal would have an immense impact on lung cancer management by enabling an early stage cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged above 21 years, capable of giving consent and suspected of lung cancer with radiological lung nodules and masses.

Exclusion Criteria:

* Patients with contra-indications to bronchoscopy and CT-TTNA that include active myocardial ischemia, uncorrected coagulopathy, severe respiratory distress, uncontrollable cough, and pregnancy will be excluded. Before females in the reproductive age are recruited, urine pregnancy test will be performed and confirmed negative.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Identification of signature VOCs as ling cancer biomarkers by comparing VOC contents between alveolar gas from lung nodules and exhaled gas.

CONTACTS AND LOCATIONS:
Overall Officials: Pyng Lee, MD, Principal Investigator — National University Hospital, Singapore; Mi Kyoung Park, Ph.D, Principal Investigator — Institute of Microelectronics
Locations (2):
- Singapore (2):
  - Institute of Microelectronics, Singapore, Singapore
  - National University Hospital/ National University of Singapore, Singapore, Singapore

REFERENCES:
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] International Early Lung Cancer Action Program Investigators; Henschke CI, Yankelevitz DF, Libby DM, Pasmantier MW, Smith JP, Miettinen OS. Survival of patients with stage I lung cancer detected on CT screening. N Engl J Med. 2006 Oct 26;355(17):1763-71. doi: 10.1056/NEJMoa060476. PMID 17065637
- [Background] Sit AK, Sihoe AD, Suen WS, Cheng LC. Positron-emission tomography for lung cancer in a tuberculosis-endemic region. Asian Cardiovasc Thorac Ann. 2010 Feb;18(1):33-8. doi: 10.1177/0218492309352119. PMID 20124294
- [Background] Mahadevia PJ, Fleisher LA, Frick KD, Eng J, Goodman SN, Powe NR. Lung cancer screening with helical computed tomography in older adult smokers: a decision and cost-effectiveness analysis. JAMA. 2003 Jan 15;289(3):313-22. doi: 10.1001/jama.289.3.313. PMID 12525232
- [Background] Phillips M, Gleeson K, Hughes JM, Greenberg J, Cataneo RN, Baker L, McVay WP. Volatile organic compounds in breath as markers of lung cancer: a cross-sectional study. Lancet. 1999 Jun 5;353(9168):1930-3. doi: 10.1016/S0140-6736(98)07552-7. PMID 10371572
- [Background] Phillips M, Cataneo RN, Cummin AR, Gagliardi AJ, Gleeson K, Greenberg J, Maxfield RA, Rom WN. Detection of lung cancer with volatile markers in the breath. Chest. 2003 Jun;123(6):2115-23. doi: 10.1378/chest.123.6.2115. PMID 12796197
- [Background] Mazzone PJ. Analysis of volatile organic compounds in the exhaled breath for the diagnosis of lung cancer. J Thorac Oncol. 2008 Jul;3(7):774-80. doi: 10.1097/JTO.0b013e31817c7439. PMID 18594325
- [Background] Filipiak W, Sponring A, Mikoviny T, Ager C, Schubert J, Miekisch W, Amann A, Troppmair J. Release of volatile organic compounds (VOCs) from the lung cancer cell line CALU-1 in vitro. Cancer Cell Int. 2008 Nov 24;8:17. doi: 10.1186/1475-2867-8-17. PMID 19025629
- [Background] Phillips M, Altorki N, Austin JH, Cameron RB, Cataneo RN, Greenberg J, Kloss R, Maxfield RA, Munawar MI, Pass HI, Rashid A, Rom WN, Schmitt P. Prediction of lung cancer using volatile biomarkers in breath. Cancer Biomark. 2007;3(2):95-109. doi: 10.3233/cbm-2007-3204. PMID 17522431
- [Background] Di Natale C, Macagnano A, Martinelli E, Paolesse R, D'Arcangelo G, Roscioni C, Finazzi-Agro A, D'Amico A. Lung cancer identification by the analysis of breath by means of an array of non-selective gas sensors. Biosens Bioelectron. 2003 Sep;18(10):1209-18. doi: 10.1016/s0956-5663(03)00086-1. PMID 12835038
- [Background] Mazzone PJ, Hammel J, Dweik R, Na J, Czich C, Laskowski D, Mekhail T. Diagnosis of lung cancer by the analysis of exhaled breath with a colorimetric sensor array. Thorax. 2007 Jul;62(7):565-8. doi: 10.1136/thx.2006.072892. Epub 2007 Feb 27. PMID 17327260
- [Background] Peng G, Trock E, Haick H. Detecting simulated patterns of lung cancer biomarkers by random network of single-walled carbon nanotubes coated with nonpolymeric organic materials. Nano Lett. 2008 Nov;8(11):3631-5. doi: 10.1021/nl801577u. Epub 2008 Oct 8. PMID 18839997
- [Background] Machado RF, Laskowski D, Deffenderfer O, Burch T, Zheng S, Mazzone PJ, Mekhail T, Jennings C, Stoller JK, Pyle J, Duncan J, Dweik RA, Erzurum SC. Detection of lung cancer by sensor array analyses of exhaled breath. Am J Respir Crit Care Med. 2005 Jun 1;171(11):1286-91. doi: 10.1164/rccm.200409-1184OC. Epub 2005 Mar 4. PMID 15750044
- [Background] Peng G, Tisch U, Adams O, Hakim M, Shehada N, Broza YY, Billan S, Abdah-Bortnyak R, Kuten A, Haick H. Diagnosing lung cancer in exhaled breath using gold nanoparticles. Nat Nanotechnol. 2009 Oct;4(10):669-73. doi: 10.1038/nnano.2009.235. Epub 2009 Aug 30. PMID 19809459
- [Background] Carlborg CF, Gylfason KB, Kazmierczak A, Dortu F, Banuls Polo MJ, Maquieira Catala A, Kresbach GM, Sohlstrom H, Moh T, Vivien L, Popplewell J, Ronan G, Barrios CA, Stemme G, van der Wijngaart W. A packaged optical slot-waveguide ring resonator sensor array for multiplex label-free assays in labs-on-chips. Lab Chip. 2010 Feb 7;10(3):281-90. doi: 10.1039/b914183a. Epub 2009 Nov 12. PMID 20090999